CLINICAL TRIAL: NCT06061588
Title: Potential Effects of Virtual Reality Technology on the Treatment of Migraine-Type Headaches: Randomized Observational Study
Brief Title: "Potential Effects of Virtual Reality Technology on the Treatment of Migraine-Type Headaches"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Safa Dönmez, M.D., Ankara City Hospital Bilkent
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Virtual Reality in Migraine
Record Dates: First submitted 2023-09-23; First posted 2023-09-29 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Migraine Disorders; Virtual Reality
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Intervention Model Description: The study is planned to be conducted at two centers. Patients visiting one hospital will receive standard treatment, while patients visiting the other hospital will receive standard treatment plus VR goggles as part of their therapy. The group receiving standard treatment will constitute the case group, while the other group will form the control group.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The case group (No Intervention): Included in the case group, patients diagnosed with migraine and experiencing headache will receive standard treatment, consisting of 50 mg of dexketoprofen within 150 cc of normal saline.
- The control group (Experimental): The control group, in addition to standard treatment, will be treated with virtual reality therapy using VR goggles, which will create a virtual environment simulating moonlight by the dark seaside or a campfire ambiance with classical music (calm, slow, and soothing).
  Interventions: Device: Virtual Reality

INTERVENTIONS:
Device: Virtual Reality — The use of virtual reality as an adjunct to routine treatment.
  Arms: The control group

SUMMARY:
The primary objective of this research is to investigate the effects of virtual reality technology on the treatment of migraine-type headaches and assess how this technology may impact the severity, frequency, and duration of headaches.

DETAILED DESCRIPTION:
This is a non-randomized controlled prospective study with the primary objective of investigating the effects of virtual reality technology on the treatment of migraine-type headaches and assessing how this technology can potentially influence the severity, frequency, and duration of headaches. Additionally, the study aims to analyze the impact of virtual reality technology on the neurological and psychological components of headaches, evaluate potential improvements in the quality of life for migraine patients undergoing virtual reality therapy, monitor the long-term effects of virtual reality in migraine treatment, and assess its sustainability. The study is divided into two arms, labeled as Arm 1 and Arm 2, with randomization being carried out by the principal investigator. All patients consenting to participate in the study will receive a standard treatment of 150 cc normal saline containing arveles (50 mg dexketoprofen), and no patient will be left untreated. One group will receive only the standard treatment (control group), while the other group will receive both the standard treatment and, in addition, virtual reality therapy consisting of a virtual environment simulating moonlight by the dark seaside or a campfire ambiance with classical music (calm, slow, and soothing) using virtual reality goggles.

Prior to medication administration (0.min) and at 15, 30, 60, and 120 minutes, patients' VAS scores will be recorded. Adult patients diagnosed with migraines who have agreed to participate in the study will be included. Patients will be eligible to participate in the study if they meet specific inclusion criteria. The severity of pain in patients diagnosed with migraines and the effectiveness of treatments used for migraine attacks will constitute the dependent variables of the study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Under the age of 65
* Willing to participate in the study
* Previously diagnosed with migraine
* Marking a VAS score of 50 or higher
* Not considered for any additional preliminary diagnosis
* No known adverse history to the active ingredient of the medication to be used
* Conscious
* Cooperatively oriented

Exclusion Criteria:

* Under 18 years of age or over 65 years of age
* Not willing to participate in the study
* Displaying vital signs outside of normal limits
* With a known history of adverse reactions to NSAIDs
* Unable to determine the severity of pain on the VAS
* Scoring 50 mm or lower on the VAS
* Pregnant individuals
* Individuals with advanced systemic illness
* Those with malignancies
* Patients with chronic liver and kidney disease
* Using sedative and analgesic neuro-psychiatric drugs
* With a history of psychological and neurological diseases
* Having taken analgesics within 8 hours prior to examination

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-03-10 (Actual); Study Completion 2024-03-10 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 0. -15. -30.-60.-120. minutes
  The change in patients' pain conditions with treatment. The pain is determined using a 100 mm scale. Patients are instructed to mark the level of pain they experience, with 0 mm indicating no pain and 100 mm indicating the presence of maximum pain.
Rescue analgesic use | 120.minute
  For patients with a VAS score 50mm or higher at 120.minute rescue therapy was planned.

SECONDARY OUTCOMES:
Side effects | 120.minute
  The difference between two groups observed in terms of side effects were recorded.

CONTACTS AND LOCATIONS:
Overall Officials: SAFA DÖNMEZ, M.D., Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bagher SM, Felemban OM, Alandijani AA, Tashkandi MM, Bhadila GY, Bagher AM. The effect of virtual reality distraction on anxiety level during dental treatment among anxious pediatric patients: a randomized clinical trial. J Clin Pediatr Dent. 2023 Jul;47(4):63-71. doi: 10.22514/jocpd.2023.036. Epub 2023 Jul 3. PMID 37408348
- [Background] Almedhesh SA, Elgzar WT, Ibrahim HA, Osman HA. The effect of virtual reality on anxiety, stress, and hemodynamic parameters during cesarean section: A randomized controlled clinical trial. Saudi Med J. 2022 Apr;43(4):360-369. doi: 10.15537/smj.2022.43.4.20210921. PMID 35414614
- [Background] Genc H, Korkmaz M, Akkurt A. The Effect of Virtual Reality Glasses and Stress Balls on Pain and Vital Findings During Transrectal Prostate Biopsy: A Randomized Controlled Trial. J Perianesth Nurs. 2022 Jun;37(3):344-350. doi: 10.1016/j.jopan.2021.09.006. Epub 2022 Apr 7. PMID 35397973
- [Background] Stepien A, Kozubski W. [Comparison of the effectiveness of lysine acetylsalicylate and metoclopramide combination with ergotamine plus caffeine in the treatment of migraine attacks]. Wiad Lek. 2004;57(3-4):135-9. Polish. PMID 15307520
- [Background] Chabriat H, Joire JE, Danchot J, Grippon P, Bousser MG. Combined oral lysine acetylsalicylate and metoclopramide in the acute treatment of migraine: a multicentre double-blind placebo-controlled study. Cephalalgia. 1994 Aug;14(4):297-300. doi: 10.1046/j.1468-2982.1994.1404297.x. PMID 7954760
- [Background] Yavuz E, Gulacti U, Lok U, Turgut K. Intravenous metoclopramide versus dexketoprofen trometamol versus metoclopramide+ dexketoprofen trometamol in acute migraine attack in the emergency department: A randomized double-blind controlled trial. Am J Emerg Med. 2020 Nov;38(11):2254-2258. doi: 10.1016/j.ajem.2020.04.038. Epub 2020 Apr 15. PMID 32359776